CLINICAL TRIAL: NCT00786201
Title: A Phase 2, Multicenter, Multinational, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-ranging Study Evaluating the Efficacy and Safety of CNTO 888 Administered Intravenously in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: A Study to Evaluate the Safety and Effectiveness of CNTO 888 Administered Intravenously (IV) in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR015235; CNTO888PUL2001 (Other: Centocor)
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-11

CONDITIONS: Pulmonary Fibrosis
Keywords: CNTO 888; Idiopathic Pulmonary Fibrosis; IPF
MeSH Terms: conditions — Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis | interventions — carlumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CNTO 888 1 mg/kg (Experimental)
  Interventions: Drug: CNTO 888 1 mg/kg
- CNTO 888 5 mg/kg (Experimental)
  Interventions: Drug: CNTO 888 5 mg/kg
- CNTO 888 15 mg/kg (Experimental)
  Interventions: Drug: CNTO 888 15 mg/kg

INTERVENTIONS:
Drug: Placebo — Intravenous (IV) infusion every 4 weeks, from Week 0 through Week 48
  Arms: Placebo
Drug: CNTO 888 1 mg/kg — IV infusion every 4 weeks, from Week 0 through Week 48
  Arms: CNTO 888 1 mg/kg
Drug: CNTO 888 5 mg/kg — IV infusion every 4 weeks, from Week 0 through Week 48
  Arms: CNTO 888 5 mg/kg
Drug: CNTO 888 15 mg/kg — IV infusion every 4 weeks, from Week 0 through Week 48
  Arms: CNTO 888 15 mg/kg

SUMMARY:
The experimental drug CNTO 888 is currently being studied in cancer patients with solid tumors and this study is the first to use this drug for patients with idiopathic pulmonary fibrosis (IPF). This study tests the safety and effectiveness of CNTO 888 compared to placebo. The purpose of this research study is to determine if CNTO 888 is safe and to determine its effects (good and bad) on patients with IPF. The study will be conducted at approximately 28 sites globally. Patients can remain on usual, accepted treatment for IPF while enrolled in the study. Participating in other experimental studies or taking other experimental medications while participating in this study will not be allowed.

DETAILED DESCRIPTION:
This study tests the safety and effectiveness of an experimental drug, CNTO 888, compared to placebo. The purpose of this research study is to determine if CNTO 888 is safe and to determine its effects on patients with idiopathic pulmonary fibrosis (IPF). CNTO 888 has not been approved by any regulatory authority for use in patients with any condition. The screening phase of the study, where the study doctor will determine if a patient is eligible for the study will last for 1 to 4 weeks. The study will enroll and treat the first 20 patients as part of a safety evaluation, at selected sites. The patients will be randomized to placebo or 1 mg/kg or 5 mg/kg or 15 mg/kg CNTO 888. The study drug will be given through a needle inserted into the patient's vein (IV). A Data Monitoring Committee will be responsible to review this portion of the study, and the study in general. They will review all of the information from patients in this portion of the study, after patients have received three infusions of study agent, or 3 months have passed since the first patient was enrolled. After their review, they will recommend whether to continue enrolling additional patients for the remainder of the study, or require some modification to the study. Patients will receive study agent until Week 48 and will continue to be followed through Week 72 for assessment of safety and any other effects after discontinuation of therapy. Patients will be in the study for about 74 weeks. The end of the study is defined as the last visit of the last patient. Patients will be randomly assigned to 1 of 4 treatment groups. Group 1, placebo IV infusion administered over 90 minutes every 4 weeks, from Week 0 through Week 48. Group 2, CNTO 888 1 mg/kg IV infusion administered over 90 minutes every 4 weeks, from Week 0 through Week 48. Group 3, CNTO 888 5 mg/kg IV infusion administered over 90 minutes every 4 weeks, from Week 0 through Week 48. Group 4, CNTO 888 15 mg/kg IV infusion administered over 90 minutes every 4 weeks, from Week 0 through Week 48. Enrollment completed as planned. Dosing terminated after interim DMC (Data Monitoring Committee) review. Participants followed until trial completed.

ELIGIBILITY:
Inclusion Criteria:

* Forced Vital Capacity (FVC) >= (greater than or equal to) 50% of the predicted value at screening
* Abnormal lung function test results that include evidence of restriction and impaired gas exchange, or evidence of desaturation at rest or exercise or decreased diffusing capacity of the lung for carbon monoxide (DLCO)
* Bibasilar reticular abnormalities with minimal ground-glass opacities on high-resolution computed tomography (HRCT) scans
* Have surgical lung biopsy evidence of usual interstitial pneumonia (UIP) and/or HRCT scan-based diagnosis of IPF
* Relative decrease of >= 10% in forced vital capacity (FVC), or relative decrease of >= 15% in DLCO, or evidence of clinically significant worsening on HRCT (eg, development of honeycombing, increase in opacities), or significant worsening of dyspnea at rest or with exertion.

Exclusion Criteria:

* Have evidence of interstitial pneumonia other than IPF
* Diagnosis of IPF is not confirmed by HRCT or lung biopsy results
* Partial pressure of oxygen in arterial blood (PaO2) < 55 mmHg (sea level) or 50 mmHg (altitude) at rest on room air
* Have a diagnosis of other significant respiratory disorder (eg, asthma, tuberculosis (TB), sarcoidosis, aspergillosis, chronic obstructive pulmonary disease [COPD], or cystic fibrosis)
* Have obstruction on prebronchodilator pulmonary function tests (PFTs) (defined as FEV1/FVC < 0.7) at screening or demonstrate an increase in FEV1 >= 12% postbronchodilator.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Rate of Percent Change (Relative to Baseline per 4 Week Interval) in Forced Vital Capacity (FVC) Through Week 52 | Baseline through Week 52
  The FVC is one component of pulmonary function testing, done with a spirometer.

SECONDARY OUTCOMES:
Time to Disease Progression | Baseline through Week 52
  The time to disease progression is defined as the time in days from randomization to occurrence of acute idiopathic pulmonary fibrosis (IPF) exacerbation or lung transplantation or all-cause mortality, whichever occurs first.
Absolute Change From Baseline in Forced Vital Capacity (FVC) at Week 52 | Baseline through Week 52
  The FVC is one component of pulmonary function testing, done with a spirometer.
Relative Change From Baseline in Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) at Week 52 | Baseline through Week 52
  The DLCO is a sensitive lung function parameter and is performed to determine how well oxygen passes from the air sacs of the lungs into the blood.
Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score at Week 52 | Baseline through Week 52
  The SGRQ is a 76-item questionnaire designed to measure the impact of respiratory disease and its treatment on the participants' health outcomes. The SGRQ is divided into 3 components: 1) symptoms, 2) activity limitations and 3) Impacts on social and psychological functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (30):
- United States (17):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Miami, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Wichita, Kansas
  - New Orleans, Louisiana
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Spartanburg, South Carolina
  - Nashville, Tennessee
  - Salt Lake City, Utah
  - Colchester, Vermont
- Leuven, Belgium
- Canada (6):
  - Edmonton, Alberta
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - London, Ontario
  - Vancouver
- Germany (2):
  - Bad Berka
  - Essen
- Netherlands (4):
  - Amsterdam
  - Nieuwegein
  - Rotterdam
  - Sittard

REFERENCES:
- [Result] Raghu G, Martinez FJ, Brown KK, Costabel U, Cottin V, Wells AU, Lancaster L, Gibson KF, Haddad T, Agarwal P, Mack M, Dasgupta B, Nnane IP, Flavin SK, Barnathan ES. CC-chemokine ligand 2 inhibition in idiopathic pulmonary fibrosis: a phase 2 trial of carlumab. Eur Respir J. 2015 Dec;46(6):1740-50. doi: 10.1183/13993003.01558-2014. Epub 2015 Oct 22. PMID 26493793